CLINICAL TRIAL: NCT02026544
Title: Evaluation of the Effect of Low Frequency Therapeutic Ultrasound (LOTUS) on Kidney Function in Chronic Kidney Disease
Brief Title: Effect of Low Frequency Ultrasound on Kidney Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonogenix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PRO-0001
Record Dates: First submitted 2013-12-19; First posted 2014-01-03 (Estimated); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Chronic Kidney Disease
Keywords: low frequency ultrasound; glomerular filtration rate
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Low Frequency Therapeutic Ultrasound (Experimental): Low Frequency Therapeutic Ultrasound (LOTUS) applied transcutaneously
  Interventions: Device: Low Frequency Therapeutic Ultrasound

INTERVENTIONS:
Device: Low Frequency Therapeutic Ultrasound — 29 kHz (kilohertz) low frequency therapeutic ultrasound delivered transcutaneously

SUMMARY:
The purpose of this study is to find out what effect, if any, Low Frequency Therapeutic Ultrasound (LOTUS) has on kidney function in patients with chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Must be >/= 18 years of age
* Must have documented Stage 3 to Stage 4 (eGFR 15 - 59) chronic kidney disease
* Females with childbearing potential must not be pregnant at the time of study
* Subject must provide written informed consent

Exclusion Criteria:

* Unable or unwilling to cooperate with study procedures
* Currently enrolled in another clinical study for which the follow-up period is not complete

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-01-28 (Actual); Primary Completion 2014-10-06 (Actual); Study Completion 2014-10-06 (Actual)

PRIMARY OUTCOMES:
Glomerular Filtration Rate (GFR) | Baseline and 15 minutes after start of Intervention
  Absolute change in glomerular filtration rate, GFR, measured by Tc-99m DTPA (diethylenetriamine pentaacetic acid) imaging (Gates Method) in the treated kidney(s) from baseline to during LOTUS

SECONDARY OUTCOMES:
Percent change in GFR | Baseline and 15 minutes after start of Intervention
  Percent change in GFR in the treated kidney(s) from baseline to during LOTUS.
Blood Pressure | Baseline and 15 minutes after start of Intervention, and 5 minutes after end of intervention
  Blood pressure is measured at baseline, during LOTUS intervention, and immediately after LOTUS intervention

OTHER OUTCOMES:
Cutaneous Injury | 5 minutes after LOTUS intervention
  Occurrence of cutaneous injury, such as erythema, blistering or rash occuring below the site of transducer placement
Heart rate | Baseline and 15 minutes after start of Intervention, and 5 minutes after end of intervention.
  Heart rate will be measured at baseline, during LOTUS intervention, and immediately after LOTUS intervention has ended.

CONTACTS AND LOCATIONS:
Overall Officials: Randall A Hawkins, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Department of Radiology and Biomedical Imaging, UCSF, San Francisco, California, United States

REFERENCES:
- [Result] Dae MW, Liu KD, Solomon RJ, Gao DW, Stillson CA. Effect of Low-Frequency Therapeutic Ultrasound on Induction of Nitric Oxide in CKD: Potential to Prevent Acute Kidney Injury. Kidney Dis (Basel). 2020 Nov;6(6):453-460. doi: 10.1159/000509819. Epub 2020 Aug 21. PMID 33313066